CLINICAL TRIAL: NCT05479188
Title: Comparative Analysis of the Microcirculation During Cardiac Surgery With Minimal Invasive Versus Conventional Extracorporeal Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Kyriakos Anastasiadis, Professor of Cardiac Surgery, Head of Cardiothoracic Department, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AUS_CTS
Record Dates: First submitted 2022-07-22; First posted 2022-07-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Aortic Valve Stenosis; Mitral Disease
Keywords: extracorporeal circulation; Minimal Invasive Extracorporeal Circulation; cardiopulmonary bypass; cerebral oximetry; microcirculation; near-infrared spectroscopy
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis; Disease

STUDY DESIGN:
Intervention Model Description: All eligible patients will be randomized with computer-generated algorithm to receive cardiac surgery with minimal invasive versus conventional extracorporeal circulation.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Invasive Extracorporeal Circulation (MiECC) (Active Comparator): Patients undergoing cardiac surgery with Minimal Invasive Extracorporeal Circulation.
  Interventions: Device: Cerebral oximetry; Device: Peripheral oximetry; Device: Cerebral autoregulation; Device: Sublingual microscopy
- Conventional cardiopulmonary Bypass (cCPB) (Active Comparator): Patients undergoing cardiac surgery with conventional cardiopulmonary bypass.
  Interventions: Device: Cerebral oximetry; Device: Peripheral oximetry; Device: Cerebral autoregulation; Device: Sublingual microscopy

INTERVENTIONS:
Device: Cerebral oximetry — Cerebral oximetry monitoring with near-infrared spectroscopy.
Device: Peripheral oximetry — Tissue perfusion monitoring with somatic near-infrared spectroscopy.
Device: Cerebral autoregulation — Cerebral autoregulation monitoring with COx.
Device: Sublingual microscopy — Evaluation of microcirculation with sublingual microscopy.

SUMMARY:
The aim of the proposed study is to evaluate microcirculatory alterations in patients undergoing open heart surgery with minimal invasive versus conventional extracorporeal circulation. Positive clinical results evidenced with goal-directed perfusion and cerebral oximetry monitoring could be attributed to preserved microcirculation at tissue level.

DETAILED DESCRIPTION:
The aim of the proposed study is to evaluate microcirculatory alterations in patients undergoing open heart surgery with minimal invasive versus conventional extracorporeal circulation.

Microcirculatory changes during cardiac surgery have been investigated mainly during coronary procedures using the conventional extracorporeal circulation.There is no single study in the literature investigating microcirculatory alterations using a perioperative strategy of "physiologic" perfusion.

Positive clinical results evidenced with goal-directed perfusion and cerebral oximetry monitoring could be attributed to preserved microcirculation at tissue level.

All patients will follow the same anaesthetic and perfusion protocol. The patients will be randomized to two arms:

1. Patients operated with Minimal Invasive Extracorporeal Circulation (MiECC)
2. Patients operated with conventional cardiopulmonary bypass (cCPB)

The protocol for the evaluation of microcirculation will be based on:

* Cerebral near-infrared spectroscopy (rScO2) measurements (INVOS, Covidien-Medtronic Inc.).
* NIRS-Based Cerebral Autoregulation Monitoring: Analog arterial blood pressure signals will be digitized and then processed with the digital NIRS signals using a personal computer and a special ICM software (University of Cambridge, Cambridge, UK). Monitoring cerebral autoregulation ensures adequate renal perfusion. Hence, brain can be used not just as a target but also as an index organ indicating adequacy of perfusion.
* Somatic near-infrared spectroscopy (rSsO2) measurements (INVOS, Covidien-Medtronic Inc.).
* Sublingual mucosal microcirculation measurements during surgery using side dark field (SDF) imaging (MicroScan, Microvision Medical, Amsterdam, The Netherlands).

All measurements will be performed at the following time points:

T0: after induction of anaesthesia T1: after initiation of cardiopulmonary bypass T2: 10 minutes after cross- clamping the aorta T3: 10 minutes before removing the aortic cross-clamp T4: after weaning from extracorporeal circulation

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing undergoing open heart surgery with accepted indications under extracorporeal circulation

Exclusion Criteria:

* patients undergoing emergency surgery
* patients in preoperative cardiogenic shock with evidence of tissue malperfusion
* patients with severe peripheral vascular disease
* patients unable to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of perfused vessels assessed with sublingual microscopy | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Proportion of perfused vessels (PPV) assessed with sublingual microscopy.
Total vessel density assessed with sublingual microscopy | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Total vessel density (TVD) assessed with sublingual microscopy.
Perfused vessel density assessed with sublingual microscopy | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Perfused vessel density (PVD) assessed with sublingual microscopy.

SECONDARY OUTCOMES:
Cerebral oximetry | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Change in cerebral oxygen saturation during cardiac surgery assessed with near-infrared spectroscopy
Peripheral tissue oximetry | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Change in tissue perfusion during cardiac surgery assessed with near-infrared spectroscopy
Cox index assessed with near-infrared spectroscopy | During surgery, from induction of anesthesia to weaning of extracorporeal circulation
  Evaluation of cerebral autoregulation during cardiac surgery with continuous monitoring of Cox index (ICM+ software, Cambridge, UK).

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Anastasiadis, Prof., Study Director — Aristotle University Of Thessaloniki; Helena Argiriadou, Assoc. Prof., Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Cardiothoracic Department, AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anastasiadis K, Antonitsis P, Deliopoulos A, Argiriadou H. A multidisciplinary perioperative strategy for attaining "more physiologic" cardiac surgery. Perfusion. 2017 Sep;32(6):446-453. doi: 10.1177/0267659117700488. Epub 2017 Mar 10. PMID 28692337
- [Background] Yuruk K, Bezemer R, Euser M, Milstein DM, de Geus HH, Scholten EW, de Mol BA, Ince C. The effects of conventional extracorporeal circulation versus miniaturized extracorporeal circulation on microcirculation during cardiopulmonary bypass-assisted coronary artery bypass graft surgery. Interact Cardiovasc Thorac Surg. 2012 Sep;15(3):364-70. doi: 10.1093/icvts/ivs271. Epub 2012 Jun 14. PMID 22700685
- [Background] Donndorf P, Kuhn F, Vollmar B, Rosner J, Liebold A, Gierer P, Steinhoff G, Kaminski A. Comparing microvascular alterations during minimal extracorporeal circulation and conventional cardiopulmonary bypass in coronary artery bypass graft surgery: a prospective, randomized study. J Thorac Cardiovasc Surg. 2012 Sep;144(3):677-83. doi: 10.1016/j.jtcvs.2012.05.037. Epub 2012 Jun 12. PMID 22698563
- [Background] Koning NJ, Vonk AB, Meesters MI, Oomens T, Verkaik M, Jansen EK, Baufreton C, Boer C. Microcirculatory perfusion is preserved during off-pump but not on-pump cardiac surgery. J Cardiothorac Vasc Anesth. 2014 Apr;28(2):336-41. doi: 10.1053/j.jvca.2013.05.026. Epub 2013 Oct 23. PMID 24161555
- [Background] Kara A, Akin S, Ince C. The response of the microcirculation to cardiac surgery. Curr Opin Anaesthesiol. 2016 Feb;29(1):85-93. doi: 10.1097/ACO.0000000000000280. PMID 26658179